CLINICAL TRIAL: NCT01326819
Title: Comparison Study of Three Regional Oxygen Saturation (rSO2) Systems Across a Wide Range of Skin Colors
Brief Title: Comparison of Normal Readings and Repeatability Across Skin Colors
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP1962
Record Dates: First submitted 2011-03-03; First posted 2011-03-31 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2012-11

CONDITIONS: Near Infrared Spectroscopy
Keywords: Near infrared spectroscopy; Skin pigmentation; Regional oxygen saturation
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational comparison study of three commercially available regional oxygen saturation devices on a wide range of skin colors.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* of any race or ethnicity
* greater than eighteen years of age
* weighs greater than or equal to 40 kilograms
* is not currently admitted to the hospital
* is not known to be pregnant
* understands English
* is willing and able to provide informed consent and comply with study procedures

Exclusion Criteria:

* is less than eighteen years of age
* weighs less than 40 kilograms
* if known to be pregnant
* is a current patient in the hospital
* does not understand English
* has known anemia
* is unwilling and able to provide informed consent and comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The mean and standard deviation of readings with all four regional oxygen saturation devices. | Data analysis will be performed when 240 subjects have been enrolled (7 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Belani, MD, Principal Investigator — Univeristy of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States